CLINICAL TRIAL: NCT01020669
Title: Prenatal Drug Exposure: Effects on the Adolescent Brain and Behavior Development: Supplementary Control Subjects Recruitment
Brief Title: Prenatal Drug Exposure: Effects on the Adolescent Brain and Behavior Development
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910455; 10-DA-N455
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-07-13

CONDITIONS: Drug Abuse; Prenatal Drug Exposure
Keywords: fMRI; Prenatal Drug Exposure; Decision Making; Working Memory; Vulnerability
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Recent research has suggested that prenatal exposure to drugs may affect specific brain processes, including working memory, stress response, and decision making. However, most of the research on the effects of prenatal drug exposure in humans has been conducted early in life, and very little is known about effects of prenatal drug exposure during the crucial brain development period that takes place during puberty and adolescence. The biological and psychological changes associated with puberty may increase adolescents' sensitivity to prenatal substance exposure. Researchers are interested in using functional magnetic resonance imaging (fMRI) scans to study brain function and learn more about the effects of prenatal drug exposure on adolescents.

Objectives:

- To examine the effects of prenatal substance exposure on working memory, decision making, and normal brain activity in adolescents.

Eligibility:

- Adolescents between 12 and 17 years of age who are enrolled in a larger follow-up study of children exposed to drugs in utero.

Design:

* The study will involve a single outpatient session with two fMRI scans that will test working memory and decision-making processes.
* Participants will have brief medical history, a physical examination, and a urine test for drugs of abuse.
* Participants will then be trained on the working memory and decision-making tasks before having an initial MRI scan to provide a baseline reading.
* The fMRI scans will take 40 to 45 minutes each, and participants will have break in between as needed.

DETAILED DESCRIPTION:
Objective- To use fMRI to compare brain activity at rest and during working memory and decision making tasks in normal children and in children exposed in utero to drugs of abuse.

Study population- All participants will be 12-17 year-olds enrolled in an ongoing longitudinal follow up study of children exposed to drugs of abuse in utero funded by NIH. A subgroup of this study cohort will be invited to participate based on added criteria needed for scanning studies, such as absence of metal in the body, no significant CNS disease, and ability to tolerate the scanning environment.

Design- Participants will undergo fMRI scans while performing a working memory task, a decision making task and at rest. Data from participants in the current study will be combined with those from a previous study (NIDA protocol 417) which now reside in our repository protocol, 8002.

Outcome measures- The primary outcome measures will be the difference in BOLD fMRI activation between drug-exposed participants and those without prenatal exposure to drugs of abuse.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participants must be enrolled in the current UMB longitudinal study protocol.
  2. All participants will be between 12 and 17 years old (inclusive).
  3. All participants must be able to provide informed assent and have a parent/guardian who can provide informed consent.

EXCLUSION CRITERIA:

1. Report of a history of significant medical/neurological illness that might interfere with imaging data such as HIV positive status, cerebral vascular accident (CVA), central nervous system (CNS) tumor, head trauma, multiple sclerosis (MS) or other demyelinating diseases, epilepsy, or movement disorders.
2. Metallic devices in the body that preclude MRI scanning, as determined by self and parent (guardian) report.
3. Current use of psychotropic medication that may alter attentional functioning (e.g., Clonidine, antipsychotics, Effexor, stimulants).
4. Currently using respiratory, cardiovascular, anticonvulsant or other medications that might interfere with the mechanisms producing the BOLD signal.
5. Currently abusing street drugs as assessed by history and urine testing.
6. Pregnancy, which will be assessed by history during screening and by urine testing on scan days.
7. Claustrophobia by self and/or parent (guardian) report severe enough to preclude toleration of the scanning environment.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2009-10-16; Study Completion 2011-07-13

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland at Baltimore/MPRC, Catonsville, Maryland, United States

REFERENCES:
- [Background] Accornero VH, Morrow CE, Bandstra ES, Johnson AL, Anthony JC. Behavioral outcome of preschoolers exposed prenatally to cocaine: role of maternal behavioral health. J Pediatr Psychol. 2002 Apr-May;27(3):259-69. doi: 10.1093/jpepsy/27.3.259. PMID 11909933
- [Background] Bandstra ES, Morrow CE, Anthony JC, Accornero VH, Fried PA. Longitudinal investigation of task persistence and sustained attention in children with prenatal cocaine exposure. Neurotoxicol Teratol. 2001 Nov-Dec;23(6):545-59. doi: 10.1016/s0892-0362(01)00181-7. PMID 11792524
- [Background] Ashtari M, Kumra S, Bhaskar SL, Clarke T, Thaden E, Cervellione KL, Rhinewine J, Kane JM, Adesman A, Milanaik R, Maytal J, Diamond A, Szeszko P, Ardekani BA. Attention-deficit/hyperactivity disorder: a preliminary diffusion tensor imaging study. Biol Psychiatry. 2005 Mar 1;57(5):448-55. doi: 10.1016/j.biopsych.2004.11.047. PMID 15737658